CLINICAL TRIAL: NCT01917539
Title: Efficacy of Pulsed Light Therapy for Meibomian Gland Dysfunction and Dry Eye Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trouble enrolling patients
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dr. Wendy Lee, Associate Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120140
Record Dates: First submitted 2013-07-19; First posted 2013-08-06 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Syndrome
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Treatment (Sham Comparator): Sham light treatment will consist of applying the usual eye shields used for PLT, applying the usual skin gel to the facial region, and applying the cooling probe without application of pulsed light therapy treatment. All subjects will come for their initial visit where evaluation and treatment #1 will take place. They will also attend 3 follow-up visits spaced approximately 3-4 weeks apart during which they will have subsequent treatments and/or evaluations for their dry eyes. The visit duration will range from approximately 60-90 minutes per clinic visit.
  Interventions: Device: Sham Treatment
- Pulsed Light Therapy (Experimental): All subjects will come for their initial visit where evaluation and treatment #1 will take place. They will also attend 3 follow-up visits spaced approximately 3-4 weeks apart during which they will have subsequent treatments and/or evaluations for their dry eyes. The visit duration will range from approximately 60-90 minutes per clinic visit.
  Interventions: Device: Pulsed Light Therapy

INTERVENTIONS:
Device: Sham Treatment — Sham light treatment will consist of applying the usual eye shields used for PLT, applying the usual skin gel to the facial region, and applying the cooling probe without application of pulsed light therapy treatment.
  Arms: Sham Treatment
Device: Pulsed Light Therapy — Light treatment will consist of applying eye shields used for PLT, applying the skin gel to the facial region, and applying the probe with application of pulsed light therapy treatment.
  Arms: Pulsed Light Therapy

SUMMARY:
Our primary aim is to determine whether pulsed light therapy (PLT) is effective in reducing symptoms and improving clinical stigmata of dry eye syndrome (DES) associated with meibomian gland dysfunction (MGD) in patients with facial rosacea (which includes ocular rosacea). The uses of PLT are for treatment of rosacea, hair removal, pigmented lesions, and skin telangiectasias. The risks include the potential for transient sunburn-like sensations (i.e. redness, burning sensation) and particularly if not used properly, the potential to cause burns, blistering, scarring, and pigmentary changes.

DETAILED DESCRIPTION:
Group 1: pre-existing dry eye treatment regimen + sham light treatment. Sham light treatment will consist of applying the usual eye shields used for PLT, applying the usual skin gel to the facial region, and applying the cooling probe without application of pulsed light therapy treatment.

Group 2: pre-existing dry eye treatment regimen + pulsed light therapy (PLT)

Subjects will be recruited from the outpatient clinics at Bascom Palmer Eye Institute, will have a chief complaint of dry eyes, and will have to meet all inclusion/exclusion criteria. Subjects will be randomized via computerassisted random number generation to Group 1 or 2. All subjects will undergo baseline evaluation for DES including a standardized questionnaire about symptoms of dry eyes (takes about 5 minutes to complete and assesses the presence and severity of dry eye symptoms), various testing on the properties and composition of the tear film, grading of changes related to dry eye seen on the surface of the eye, and grading of the oil glands on the eyelid (meibomian glands) and their secretions. Primary outcomes will be anatomical improvement of the meibomian glands and their secretions.

Subjects in Group 1 will continue their pre-existing dry eye treatment regimen and receive sham light treatment, whereas subjects in Group 2 will continue their pre-existing dry eye treatment regimen and receive PLT. All subjects will come for their initial visit where evaluation and treatment #1 will take place. They will also attend 3 follow-up visits spaced approximately 3-4 weeks apart during which they will have subsequent treatments and/or evaluations for their dry eyes. The visit duration will range from approximately 60-90 minutes per clinic visit.

The PLT devices are FDA approved for the treatment of rosacea in the periocular/facial region, and having facial rosacea is one of the inclusion criteria for this study. This is the indication for treatment with PLT. The devices are not FDA-approved for the treatment of DES, although this is something we will be looking at as one of our main outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 y/o
* Patients presenting to academic referral center for DES
* Diagnosis of mild to moderate DES with meibomian gland dysfunction and ocular rosacea, based on evaluation of meibomian glands (MG), MG secretions, and other factors
* Facial rosacea
* Patients must not have started any new medications within the past 1 month
* Patients should not be using warm compresses or lid scrubs more than 1-2 times in the previous 2 weeks
* Symptomatic changes in DES

Exclusion Criteria:

* Age < 18
* History of inflammatory DES (e.g. Sjogren's, rheumatoid arthritis, Stevens-Johnson syndrome, ocular cicatricial pemphigoid)
* History of trauma-induced ocular surface disease (thermal burns, chemical burns)
* Severe DES
* Pregnant women
* H/o seizures
* Significant unprotected sun exposure or use of tanning beds or creams in treated area (must be discontinued at least 2 weeks prior to treatment, during treatment course, and 2 weeks after last treatment)
* Use of Accutane, anti-coagulants, or St. John's Wort
* Active infections/immunosuppression
* Herpes 1 or 2 within the treatment area
* Patients who have undergone LASIK surgery within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Anatomical improvement of the meibomian glands and their secretions. | 3 months
  We are looking at subjective changes in DES symptomatology based on the OSDI questionnaire score. We are also looking at objective changes in examination findings based on the tear film properties (TBUT, Schirmer), staining patterns of the ocular surface using fluor. and LG dyes, characteristics of the meibomian glands and lid margin (e.g. telangiectasias, notching, myelography by transillumination, etc), as well as the meibum secretions (e.g. expressibility, and consistency).
  Change in baseline for OSDI, TBUT in seconds, Schirmer testing in mm, staining pattern score (standardized proprietary score on a scale of 1-4), myelography by % of meibomian glands that can be transilluminated, expressibility/consistency (proprietary score on scale of 1-4) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lee, MD, Principal Investigator — University of Miami Bascom Palmer Eye Institute
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Miami, Florida, United States